CLINICAL TRIAL: NCT04940013
Title: Assessing the Acceptability of Using Misoprostol Alone for Menstrual Regulation
Brief Title: Missed Period Pill Study
Acronym: MPP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of successful recruitment and loss of funding
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-30048
Record Dates: First submitted 2021-06-11; First posted 2021-06-25 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Menstrual Regulation; Menstrual Irregularity
Keywords: late period; missed period; mensturation
MeSH Terms: conditions — Menstruation Disturbances | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study participants (Other): Study participants will be persons who have late period of up to 14 days
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Study participants are given misoprostol alone for menstrual regulation.

SUMMARY:
The Missed Period Pill Study is a prospective observational study among people who decide to use misoprostol alone for menstrual regulation.

DETAILED DESCRIPTION:
As the number of state laws restricting access to abortion increases across the country, more creative methods are needed to support individuals in achieving their reproductive goals. Misoprostol alone for people who suspect, but have not confirmed pregnancy, has the potential to fulfill this growing need. The goal of this research study is to test a traditional but underutilized framework of menstrual regulation for pregnancy loss, to "bring back" a period when it is missed. This study will aim to recruit 100 patients who have a missed period to address research questions that focus on the feasibility and acceptability of using misoprostol alone for menstrual regulation.

The study will require 1 study visit and 1 telehealth visit.

First study visit: A urine sample will be collected which will later undergo pregnancy testing. Participants will be given misoprostol along with instructions and information on what to expect. The participant will be required to return to the clinic 4 weeks later to provide another urine sample. The participant will not know the results of the first visit's pregnancy test at any point. The clinic staff member administering the participant's care will not know of the pregnancy test result while the participant is at the clinic.

Telehealth visit: The second visit will be by phone or video. The participant will conduct a pregnancy test and inform the research staff of the result. The participant will then be asked to answer questions on an online survey about their experience using misoprostol.

A variety of clinical and social science measures will be collected to assess the feasibility and acceptability of this traditional concept of menstrual regulation utilizing uterine evacuation with medications.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years old or older
* Read and speak English
* Know the date of their last menstrual period within 2 days
* Have a period that is late by up to 14 days
* Have had regular periods in the last 4-6 months
* Does not want to be pregnant; understand that if they are pregnant, the pills will end their pregnancy
* Be willing to have an abortion if the missed period pill does not work, and informed of potential for birth defects in any ongoing pregnancy
* Does not want to verify pregnancy status
* Does not have risk factors for ectopic pregnancy (history of ectopic pregnancy, recent vaginal bleeding or spotting, pelvic pain on one side, prior permanent contraception, or other tubal surgery)
* Does not have an IUD
* Does not currently use a contraceptive implant or injectable
* Does not have contraindications to misoprostol
* Agree to participate in the follow up visit/call

Exclusion Criteria:

* Participants who have contraindications to misoprostol
* Unknown date of last menstrual period
* Risk factors for ectopic pregnancy (history of ectopic pregnancy, recent vaginal bleeding or spotting, pelvic pain on one side, prior permanent contraception, or other tubal surgery)
* Irregular menses or any other condition that in the opinion of the Principal Investigator would compromise participant safety.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Interest in missed period pills | Documented at Enrollment Survey
  The proportion of the clinic-going population that may be interested in a missed period pill and accept not having their pregnancy confirmed beforehand, therefore not knowing whether they terminated a pregnancy.
Satisfaction with missed period pills | Documented at Follow-up Survey, 4 weeks after drug administration
  The proportion of participants reporting being "satisfied" or "very satisfied" with the missed period pills on a five-point Likert scale at 4 weeks.

SECONDARY OUTCOMES:
Efficacy of missed period pills | Documented at the second study visit, through study completion at around 4 weeks after drug adminstration
  The proportion of participants that successfully brought down their period, resulting in a negative pregnancy test and the return of their period.

CONTACTS AND LOCATIONS:
Overall Officials: Ushma Upadhyay, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Missed Period Pill Study Enrollment Website — https://www.periodpillstudy.org/